CLINICAL TRIAL: NCT03464916
Title: A Phase 1, Open-Label, Dose-Escalation, Pharmacokinetic, and Pharmacodynamic Study of the Safety and Efficacy of CAR2 Anti-CD38 A2 CAR-T Cells in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study to Evaluate the Safety and Efficacy of Anti-CD38 CAR-T in Relapsed or Refractory Multiple Myeloma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SOR-CART-MM-001
Record Dates: First submitted 2018-02-14; First posted 2018-03-14 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: CAR2 Anti-CD38 A2 CAR-T Cells
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: To determine DLT and MTD, the design uses a 3+3 rule-based design. Dose escalation is permitted between successive cohorts based upon a specified algorithm, using discrete dosage steps.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAR2 Anti-CD38 A2 CAR-T Cells (Experimental): Relapsed or Refractory Multiple Myeloma
  Interventions: Biological: CAR2 Anti-CD38 A2 CAR-T Cells

INTERVENTIONS:
Biological: CAR2 Anti-CD38 A2 CAR-T Cells — Autologous IV infusion; dose-escalation

SUMMARY:
The study is an open-label Phase 1 single dose-escalation safety study of CAR2 Anti-CD38 A2 CAR-T Cells in patients with Relapsed or Refractory Multiple Myeloma, who meet all other eligibility criteria.

DETAILED DESCRIPTION:
All subjects who received investigational CAR-T therapy will be included in the analyses and summaries of safety, efficacy, pharmacokinetic, and pharmacodynamic assessments.

ELIGIBILITY:
Inclusion Criteria:

* The patient must either have relapsed refractory multiple myeloma (RRMM) after receiving prior lines of anti-myeloma treatments that included at least lenalidomide (Revlimid®), pomalidomide (Pomalyst®), bortezomib (Velcade®), carfilzomib (Kyprolis®), and daratumumab (Darzalex®) (refractory MM is defined as the development of disease progression during therapy with an anti-myeloma regimen or within 60 days of the last dose of an anti-myeloma regimen or the achievement of less than a partial response (PR) after greater than or equal to 2 cycles; for relapsing patients the duration from the last dose of the last prior treatment regimen to relapse must be less than or equal to 12 months); OR have multiple myeloma that is refractory to or has relapsed within 1 year of receiving high-dose therapy [HDT]/autologous stem cell transplantation [ASCT] in first- or second-line (refractory is defined as the achievement of less than a PR at the Day 90 to 100 post-ASCT response assessment)
* Must have measurable disease as defined by the following: Serum M-protein greater than or equal to 1 g/dL; OR Urine M-protein greater than or equal to 200 mg/24 hours; OR Serum free light chain (FLC) assay; involved FLC level greater than or equal to 10 mg/dL provided the serum FLC ratio is abnormal; OR greater than or equal to 30% clonal plasma cells in the bone marrow aspirate or biopsy sample
* Must have a life expectancy of at least 12 weeks
* Subjects should be willing and able to comply with the study schedule and protocols
* Females of childbearing potential must have 2 negative pregnancy tests, agree to ongoing pregnancy testing during the study, and sexually active female and male subjects must be willing to use an effective method to avoid pregnancies.

Exclusion Criteria:

* Subjects who received anticancer therapy or investigational drug within 28 days of first dose
* Subjects who received any approved anticancer chemotherapy within 21 days of first dose (exception cyclophosphamide as NMA conditioning)
* Subjects with unresolved toxicity greater than Grade 2 from previous therapies
* Have myeloma involvement of central nervous system (CNS) or a history of brain metastasis or spinal cord compression
* Subjects with an ECOG performance status greater than or equal to 3
* Has received allogenic hematopoietic stem cell transplantation (HSCT) within 6 months, have active graft-versus-host disease (GVHD) following transplant, or receiving immunosuppressive therapy following a transplant
* Has received any CAR cell line therapies
* Has any clinically significant low baseline lab results for hemoglobin, platelet counts, and neutrophil counts, at screening unless resulting from underlying RRMM.
* Has any clinically significant elevated baseline lab results for serum creatinine, AST, and total bilirubin (except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome) at screening regardless of causality.
* Known HIV or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or C.
* Female subjects who are pregnant or breastfeeding
* Active bacterial, viral or fungal infections
* Has active plasma cell leukemia
* Has medical condition, abnormality, or psychiatric illness that would prevent study participation
* Left ventricular ejection fraction (LVEF) less than 40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-08-23 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Determine the MTD | 28 days
  The MTD is assessed according to a 3+3 dose-escalation design by the occurrence of treatment-emergent dose-limiting toxicities during the 28-day Treatment Period in the dose-escalation phase of the study

SECONDARY OUTCOMES:
Determine the CAR2 Anti-CD38 A2 CAR-T cell blood concentrations (Pharmacokinetic [PK] Profile) to evaluate the Cmax | 28 days
  CAR2 Anti-CD38 A2 CAR-T cell blood concentrations will be measured at different time points during the 28-day treatment period to evaluate the maximum concentration (Cmax).
Determine the CAR2 Anti-CD38 A2 CAR-T cell blood concentrations (Pharmacokinetic [PK] Profile) to evaluate the AUC | 28 days
  CAR2 Anti-CD38 A2 CAR-T cell blood concentrations will be measured at different time points during the 28-day treatment period to evaluate the area under the curve (AUC).
Evaluate the safety of Anti-CD38 A2 CAR-T cells in Patients with RRMM by incidence of treatment-emergent adverse events | 6 months
  The evaluation of safety will be measured by an assessment of the incidence of treatment-emergent adverse events for each patient in the dose-escalation and expansion phases of the study.
Assess preliminary efficacy by response rate in accordance with the modified International Myeloma Working Group (IMWG) criteria | 6 months
  As a measure of activity, overall response rate will be assessed according to the modified International Myeloma Working Group (IMWG) criteria. Response will be assessed for each patient over a 6-month timeframe during both the dose-escalation and expansion phases of the protocol.
Assess preliminary efficacy by depth of response in accordance with the modified International Myeloma Working Group (IMWG) criteria. | 6 months
  As a measure of activity, depth of response (ie, category of response) will be assessed according to the modified International Myeloma Working Group (IMWG) criteria. This will be assessed for each patient over a 6-month timeframe during both the dose-escalation and expansion phases of the protocol.
Assess preliminary efficacy by duration of response in accordance with the modified International Myeloma Working Group (IMWG) criteria. | 6 months
  As a measure of activity, duration of response will be assessed according to the modified International Myeloma Working Group (IMWG) criteria. This will be assessed for each patient over a 6-month timeframe during both the dose-escalation and expansion phases of the protocol.
Assess preliminary efficacy by progression-free survival. | 6 months
  As a measure of activity, Progression-free survival (PFS) will be assessed. The events for the assessment of PFS are disease progression and death events. This time to event endpoint will be estimated using Kaplan-Meier methods. Point estimates and 95% confidence intervals will be provided where appropriate.
Assess preliminary efficacy by overall survival. | 6 months
  As a measure of activity, Overall Survival (OS) will be assessed. The events for the assessment of OS are death events. Time to event endpoints will be estimated using Kaplan-Meier methods. Point estimates and 95% confidence intervals will be provided where appropriate.
The determination of the recommended phase 2 dose (RP2D) will be based on an evaluation of treatment-emergent events. | 6 months
  The RP2D will be assessed by the incidence of treatment-emergent adverse events during the Treatment and Observation Periods.
The determination of the recommended phase 2 dose will be based on an evaluation of overall response rate. | 6 months
  The rate of response as a determination factor for the RP2D will be assessed by the incidence of responses of at least partial response according to the IMWG criteria during the Treatment and Observation Periods.
The determination of the recommended phase 2 dose (RP2D) will be based on an evaluation of depth of response. | 6 months
  The depth of response as a determination factor for the RP2D will be assessed by the IMWG categories for response according to changes from baseline in M-protein levels in serum and urine, per cent plasma cells in the bone marrow, and size (area) of soft tissue extramedullary plasmacytomas (if applicable). This will be assessed for each patient over a 6-month timeframe during both the dose-escalation and expansion phases of the protocol.
The determination of the recommended phase 2 dose (RP2D) will be based on an evaluation of duration of response. | 6 months
  The duration of response as a determination factor for the RP2D will be assessed by the IMWG criteria for disease progression following the achievement of a response of at least a partial response according to changes in M-protein levels in serum and urine, per cent plasma cells in the bone marrow, the appearance of new lytic bone lesions, and/or the development of new soft tissue extramedullary plasmacytomas during the Treatment and Observation periods.
The determination of the recommended phase 2 dose (RP2D) will be based on an evaluation of progression-free survival. | 6 months
  Progression-free survival as a determination factor for the RP2D will be assessed by the IMWG criteria for disease progression events and death events. This time to event endpoint will be estimated using Kaplan-Meier methods. Point estimates and 95% confidence intervals will be provided where appropriate. Progression-free survival will be evaluated during the Treatment and Observation Periods of the study.
The determination of the recommended phase 2 dose (RP2D) will be based on an evaluation of overall survival. | 6 months
  Overall survival as a determination factor for the RP2D will be assessed by death events that occur during the Treatment and Observation Periods. Time- to-event endpoints will be estimated using Kaplan-Meier methods. Point estimates and 95% confidence intervals will be provided where appropriate.

OTHER OUTCOMES:
An assessment of pharmacodynamics will be based on determining if there is an association of the achievement of at least a partial response with the level of Cmax of circulating CAR-T cells. | 6 months
  The Cmax of the concentration of circulating CAR2 anti-CD38 CAR-T cells will be determined during the Treatment Period for each patient. The achievement of at least a partial response for each patient will be assessed during both the Treatment and Observation Periods for each patient. An analysis to determine if a specific level of Cmax for the circulating CAR2 anti-CD38 CAR-T cells obtained during the Treatment Period is required for patients to achieve at least a partial response during the Treatment and Observation Periods.
An assessment of pharmacodynamics will be based on determining if there is an association of the achievement of at least a partial response with the AUC of circulating CAR-T cells. | 6 months
  The AUC of circulating CAR2 anti-CD38 CAR-T cells will be determined during the Treatment Period for each patient. The achievement of at least a partial response for each patient will be assessed during both the Treatment and Observation Periods for each patient. An analysis to determine if a specific value for the AUC of circulating CAR2 anti-CD38 CAR-T cells obtained during the Treatment Period is required for patients to achieve at least a partial response during the Treatment and Observation Periods.
An assessment of pharmacodynamics will be based on determining if there is an association of the incidence of at least Grade 3 cytokine release syndrome (CRS) adverse events with the level of Cmax of circulating CAR-T cells. | 6 months
  The Cmax of the concentration of circulating CAR2 anti-CD38 CAR-T cells will be determined during the Treatment Period for each patient. The incidence of CRS adverse events for each patient will be assessed during both the Treatment and Observation Periods for each patient. An analysis will be conducted to determine if there is a level of Cmax for circulating CAR2 anti-CD38 CAR-T cells obtained during the Treatment Period above which is associated with the development of at least Grade 3 CRS in patients during the Treatment and Observation Periods.
An assessment of pharmacodynamics will be based on determining if there is an association of the incidence of at least Grade 3 CRS with the AUC of circulating CAR-T cells. | 6 months
  The AUC of circulating CAR2 anti-CD38 CAR-T cells will be determined during the Treatment Period for each patient. The incidence of at least Grade 3 CRS for each patient will be assessed during both the Treatment and Observation Periods for each patient. An analysis to determine if there is a specific value for the AUC of circulating CAR2 anti-CD38 CAR-T cells obtained during the Treatment Period above which is associated with the development of at least Grade 3 CRS in patients during the Treatment and Observation Periods.
An assessment of pharmacodynamics will be based on determining if there is an association of the incidence of at least Grade 2 neurotoxicity adverse events with the level of Cmax of circulating CAR-T cells. | 6 months
  The Cmax of the concentration of circulating CAR2 anti-CD38 CAR-T cells will be determined during the Treatment Period for each patient. The incidence of neurotoxicity adverse events for each patient will be assessed during both the Treatment and Observation Periods for each patient. An analysis will be conducted to determine if there is a level of Cmax for circulating CAR2 anti-CD38 CAR-T cells obtained during the Treatment Period above which is associated with the development of at least Grade 2 neurotoxicity adverse events in patients during the Treatment and Observation Periods.
An assessment of pharmacodynamics will be based on determining if there is an association of the incidence of at least Grade 2 neurotoxicity adverse events with the AUC of circulating CAR-T cells. | 6 months
  The AUC of circulating CAR2 anti-CD38 CAR-T cells will be determined during the Treatment Period for each patient. The incidence of at least Grade 2 neurotoxicity adverse events for each patient will be assessed during both the Treatment and Observation Periods for each patient. An analysis to determine if there is a specific value for the AUC of circulating CAR2 anti-CD38 CAR-T cells obtained during the Treatment Period above which is associated with the development of at least Grade 2 neurotoxicity adverse events in patients during the Treatment and Observation Periods.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Stadtmauer, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Icahn School of Medicine, New York, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No